CLINICAL TRIAL: NCT06578767
Title: Decompression of Pudendal and Inferior Cluneal Nerves Using Robot-assisted Laparoscopy for Entrapment Neuralgias: Results After 1 Year of Follow-up (the X-DECO Study)
Brief Title: Decompression of Pudendal and Inferior Cluneal Nerves Using Robot-assisted Laparoscopy for Entrapment Neuralgias : the X-DECO Study
Acronym: X-DECO
Status: Recruiting | Type: Observational
Sponsor: UBOSGA (Other)
Responsible Party: Sponsor
Other Study IDs: CERU_2024-034
Record Dates: First submitted 2024-08-05; First posted 2024-08-29 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Pudendal Neuralgia
Keywords: pudendal; inferior cluneal; robot; surgery; decompression; neurolysis; laparoscopy
MeSH Terms: conditions — Pudendal Neuralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of our study is to evaluate the efficacy of the laparoscopic robot-assited approach after 1 year of follow-up, on pain experience, and anxiety, depression, post-traumatic stress syndrome and quality of life.

DETAILED DESCRIPTION:
Pudendal and inferior cluneal neuralgias are responsible for chronic pelvic perineal pain. The compression of both of the nerves are thought to be associated in approximately 25% of the pudendal neuralgias. The failure of the isolated pudendal decompression led in the early 2000s to the identification of an entrapment syndrome of the posterior femoral cutaneous nerve and its inferior cluneal branche around the ischial tuberosity. This subsequent neuralgia affects the posterior part of the perineum, lower buttock, and the posterior part of the thigh, without any associated neuro-vegetative symptoms, unlike in pudendal neuralgia. In case of failure of the medical treatment, the open trans-gluteal decompression was proposed as a gold standard. However, this technique remains invasive and requires a long recovery. In a previous study, the investigators demonstrated the feasibility of double decompression via a minimally invasive robot-assisted laparoscopic approach, and described a 4-step technique.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* Patients presenting a pudendal and inferior cluneal entrapment neuralgia with 5 positive"Nantes criteria", and failure of the medical treatment
* Patient having given consent after reading the information note

Exclusion Criteria:

* Absence of any "Nantes criteria",
* Patient non suitable for surgery/general anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This cohort study is a pilot study to evaluate decompression of pudendal and inferior cluneal nerves using robot-assisted laparoscopy for entrapment neuralgias
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Evaluate the efficacy of the surgical technique on pain experience related to pudendal and inferior cluneal chronic entrapment neuralgias, using a composite criteria (Numeric pain scale, time seated, PGIC score) | Pré-operatively, 2 days, 4 months, 1 year after surgery
  Numeric pain scale (0 "no pain" to 10 "maximal pain"), time seated (> 30 min,> 60min or unlimited) Patients' Global Impression of Change (PGIC) scale (1 "very hightly improved" to 7 "very hightly worsened") are combined to create a composite criteria (significant improvement to complete improvement)

SECONDARY OUTCOMES:
Report all complications during the follow-up | 2 days, 4 months, 1 year after surgery
  Complications are evaluated with Clavien-Dindo classification (Grade I to V(death))
Evaluate the effect of the surgical technique on anxiety | Pré-operatively, 2 days, 4 months, 1 year after surgery
  Anxiety is evaluated with STAI (State Trait Anxiety Inventory-form) (anxious personality since STAI score 51 for women, and score 61 for men)
Evaluate the effect of the surgical technique on depression | Pré-operatively, 2 days, 4 months, 1 year after surgery
  Depression is evaluated with Beck inventory (mild to moderate depression since score 10, moderate depression since score 19, severe depression since score 30)
Evaluate the effect of the surgical technique on post-traumatic stress syndrome | Pré-operatively, 2 days, 4 months, 1 year after surgery
  Post-traumatic stress syndrome is evaluated with PCL-5 (post-traumatic stress disorder checklist with a PTSD since score 38
Evaluate the impact on quality of life | Pré-operatively, 2 days, 4 months, 1 year after surgery
  Quality of life is evaluated with SF-36 (36-item Short Form Health Survey)

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Celhay, M.D, Principal Investigator — UBOSGA
Locations (1):
- UBOSGA, Bordeaux, Gironde, France